CLINICAL TRIAL: NCT03120078
Title: Diagnostic Accuracy of Ultrasound for Adenomyosis, Development of Scoring System and Correlation With Various Pelvic Pathologies: a Prospective Study.
Brief Title: A Prospective Study of Diagnostic Accuracy of Ultrasound
Status: Terminated | Type: Observational
Why Stopped: The PI has requested to close this study.
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Sushila Arya, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E17057
Record Dates: First submitted 2017-04-13; First posted 2017-04-19 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Adenomyosis
Keywords: Ultrasound
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospectively-Patients undergoing a hysterectomy for abnormal uterine bleeding (AUB) or pelvic pain will be enrolled in the study, will get pelvic ultrasound at the ultrasound clinic. An ultrasound will be obtained as part of the required clinical assessment before the patient undergoes a hysterectomy. The ultrasound images will be reviewed using Viewpoint reporting system-various sonographic features of adenomyosis will be reported detailed, including pelvic pathology, pelvic congestion syndrome etc. The histopathological examination will be done by assigned pathologist for accurate mapping/localizing the adenomyosis (appropriate section of uterus to defining localized versus generalized adenomyosis) on all patients diagnosed with adenomyosis on ultrasound. The ultrasound will be correlated with histopathology(which is the gold standard for diagnosis of adenomyosis). Scoring system for adenomyosis based on various sonographic features/clinical symptoms and their confirmation with histopathology will be developed.

DETAILED DESCRIPTION:
The association between adenomyosis, assisted reproductive technology (ART) outcomes and pregnancy complications is well established.

Adenomyosis uteri is a common gynecologic disorder with unclear etiology, characterized by the presence of hetero- topic endometrial glands and stroma in the myometrium with adjacent smooth muscle hyperplasia, defined histopathologically. Uterine adenomyosis is relatively frequent, and the diagnosis is more often made in multiparous patients in their fourth and fifth decade of life. It has been noted in 20% to 30% of the general female population and in up to 70% of hysterectomy specimens, depending on the definition used.

Accurate diagnosis and localization of the disease is important, in particular when fertility conservation is warranted. Management options include medical therapy and surgery. Medical therapies target symptomatic relief and include oral contraceptive agents, progestin therapy including the levonorgestrel-releasing intrauterine system, danazol, gonadotropin-releasing hormone agonists, and aromatase inhibitors. More uterine sparing surgical options are investigated for treatment of adenomyoisis. Surgical management can be divided into uterine sparing options such as hysteroscopic or laparoscopic resection of focal disease, endometrial ablation, uterine artery embolization, and MRgFUS, or definitive treatment via hysterectomy. The sensitivity and specificity of MRI in diagnosing adenomyosis range from 88% to 93% and 67% to 91%, respectively. Ultrasound has limitation especially when myomas are associated with adenomyosis in 36% to 50% of cases, making MRI an ideal imaging method in that scenario. The sensitivity of ultrasound to detect adenomyosis ranges from 65% to 81%, and specificity ranges from 65% to 100%. A recent meta-analysis on the accuracy of ultrasound in the diagnosis of adenomyosis demonstrated sensitivity of 82.5% (95% confidence interval, 77.5-87.9) and specificity of 84.6% (95% confidence interval, 79.8-89.8), with a positive likelihood ratio of 4.7 (3.1-7.0) and negative likelihood ratio of 0.26 (0.18-0.39), comparable to MRI.

Adenomyosis is a heterogeneous entity and thus its sonographic appearance is also variable. The variation in the degree of invasion and the heterogeneity in the reaction of surrounding tissue account for the ultrasound findings of adenomyosis. It manifests most commonly as a diffuse disease involving the entire myometrium and commonly involves the posterior uterine wall. It can also present as a localized focal entity known as nodular adenomyosis or an adenomyomas.

Following are common sonographic features of adenomyoisis.

1. Heterogeneous Myometrium: Lack of homogeneity within the myometrium, with evidence of architectural disturbance with increased and decreased echoes. This is most predictive of adenomyosis.
2. Loss of endometrium-myometrium border: Invasion of the myometrium by the glands also obscures the normally distinct endometrium-myometrium border, making it difficult to measure. This is a layer that appears as a hypoechoic halo surrounding the endometrial layer. In the past this was obtainable only with MRI; however, with newer high-resolution ultrasound, in particular using 3D rendering, it is now possible to visualize this layer. Thickness >8 to 12 mm is associated with adenomyosis.
3. Echogenic linear striations: Invasion of the endometrial glands into the subendometrial tissue induces a hyperplastic reaction that appears as echogenic linear striations fanning out from the endometrial layer.
4. Asymmetrical Uterine wall thickening: anteroposterior asymmetry, in particular when the disease is focal.
5. Color Doppler ultrasonography can also be used to differentiate adenomyosis from leiomyomas. Random scattering of vessels or intramural signals in adenomyosis cases. In contrast, in leiomyoma cases the vessels were peripheral or outer feeding vessels.

The investigators are trying to see what are the most common sonographic features of adenomyosis.

There is no clear terminology and consensus on classification of adenomyoisis on ultrasound images. Since this is a heterogeneous condition, significantly affects reproduction and newer specific uterine sparing options warrants correct localization and subclassify the disease burden like overt adenomyoisis versus localized adenomyomas. Also recently there is evidence that adenomyoisis is a progressive disease.

Presented data will aid in development of the integrated scoring system for detection and objective assessment of adenomyosis.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years or older but 60 years or less.
* Undergoing hysterectomy for AUB or pelvic pain

Exclusion Criteria:

* known cause of AUB or pelvic pain

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Patients undergoing hysterectomy for with AUB or pelvic pain will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Develop a scoring system for adenomyosis based on various sonographic features and clinical symptoms. | Duration of Study
  Sonographic features

SECONDARY OUTCOMES:
Review the diagnostic accuracy of ultrasound with adenomyosis. | Duration of study
  Various sonographic features of adenomyosis will be reported
Prevalence of coexisting pathology. | Duration of Study
  Correlation with histopathology.
Menstrual bleeding questionnaire | Duration of Study
  Comprehensive patient reported outcome instrument for heavy menstrual bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Sushila Arya, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University Health Science Center, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No
RedCap

REFERENCES:
- [Background] Devlieger R, D'Hooghe T, Timmerman D. Uterine adenomyosis in the infertility clinic. Hum Reprod Update. 2003 Mar-Apr;9(2):139-47. doi: 10.1093/humupd/dmg010. PMID 12751776
- [Background] Azziz R. Adenomyosis: current perspectives. Obstet Gynecol Clin North Am. 1989 Mar;16(1):221-35. PMID 2664619
- [Background] Vercellini P, Ragni G, Trespidi L, Oldani S, Panazza S, Crosignani PG. Adenomyosis: a deja vu? Obstet Gynecol Surv. 1993 Dec;48(12):789-94. PMID 8309661
- [Background] Farquhar C, Brosens I. Medical and surgical management of adenomyosis. Best Pract Res Clin Obstet Gynaecol. 2006 Aug;20(4):603-16. doi: 10.1016/j.bpobgyn.2006.01.012. Epub 2006 Mar 24. PMID 16563872
- [Background] Bragheto AM, Caserta N, Bahamondes L, Petta CA. Effectiveness of the levonorgestrel-releasing intrauterine system in the treatment of adenomyosis diagnosed and monitored by magnetic resonance imaging. Contraception. 2007 Sep;76(3):195-9. doi: 10.1016/j.contraception.2007.05.091. Epub 2007 Jul 27. PMID 17707716
- [Background] Garcia L, Isaacson K. Adenomyosis: review of the literature. J Minim Invasive Gynecol. 2011 Jul-Aug;18(4):428-37. doi: 10.1016/j.jmig.2011.04.004. Epub 2011 May 31. PMID 21622029
- [Background] Dong X, Yang Z. High-intensity focused ultrasound ablation of uterine localized adenomyosis. Curr Opin Obstet Gynecol. 2010 Aug;22(4):326-30. doi: 10.1097/GCO.0b013e32833bea2e. PMID 20610999
- [Background] Horng HC, Chen CH, Chen CY, Tsui KH, Liu WM, Wang PH, Chang WH, Huang BS, Sun HD, Chang TC, Chang WC, Yen MS. Uterine-sparing surgery for adenomyosis and/or adenomyoma. Taiwan J Obstet Gynecol. 2014 Mar;53(1):3-7. doi: 10.1016/j.tjog.2014.01.001. PMID 24767637
- [Background] Fukunishi H, Funaki K, Sawada K, Yamaguchi K, Maeda T, Kaji Y. Early results of magnetic resonance-guided focused ultrasound surgery of adenomyosis: analysis of 20 cases. J Minim Invasive Gynecol. 2008 Sep-Oct;15(5):571-9. doi: 10.1016/j.jmig.2008.06.010. Epub 2008 Jul 26. PMID 18657480
- [Background] Kim MD, Kim S, Kim NK, Lee MH, Ahn EH, Kim HJ, Cho JH, Cha SH. Long-term results of uterine artery embolization for symptomatic adenomyosis. AJR Am J Roentgenol. 2007 Jan;188(1):176-81. doi: 10.2214/AJR.05.1613. PMID 17179361
- [Background] Kitamura Y, Allison SJ, Jha RC, Spies JB, Flick PA, Ascher SM. MRI of adenomyosis: changes with uterine artery embolization. AJR Am J Roentgenol. 2006 Mar;186(3):855-64. doi: 10.2214/AJR.04.1661. PMID 16498121
- [Background] Pelage JP, Jacob D, Fazel A, Namur J, Laurent A, Rymer R, Le Dref O. Midterm results of uterine artery embolization for symptomatic adenomyosis: initial experience. Radiology. 2005 Mar;234(3):948-53. doi: 10.1148/radiol.2343031697. Epub 2005 Jan 28. PMID 15681687
- [Background] Wang PH, Liu WM, Fuh JL, Cheng MH, Chao HT. Comparison of surgery alone and combined surgical-medical treatment in the management of symptomatic uterine adenomyoma. Fertil Steril. 2009 Sep;92(3):876-885. doi: 10.1016/j.fertnstert.2008.07.1744. Epub 2008 Sep 6. PMID 18774566
- [Background] Wood C. Surgical and medical treatment of adenomyosis. Hum Reprod Update. 1998 Jul-Aug;4(4):323-36. doi: 10.1093/humupd/4.4.323. PMID 9825848
- [Background] Bazot M, Cortez A, Darai E, Rouger J, Chopier J, Antoine JM, Uzan S. Ultrasonography compared with magnetic resonance imaging for the diagnosis of adenomyosis: correlation with histopathology. Hum Reprod. 2001 Nov;16(11):2427-33. doi: 10.1093/humrep/16.11.2427. PMID 11679533
- [Background] Gatti GL, Michalek H. Investigations on rapeseed oil toxicology. Arzneimittelforschung. 1975 Oct;25(10):1639-42. PMID 1243051
- [Background] Dueholm M, Lundorf E, Hansen ES, Sorensen JS, Ledertoug S, Olesen F. Magnetic resonance imaging and transvaginal ultrasonography for the diagnosis of adenomyosis. Fertil Steril. 2001 Sep;76(3):588-94. doi: 10.1016/s0015-0282(01)01962-8. PMID 11532486
- [Background] Kepkep K, Tuncay YA, Goynumer G, Tutal E. Transvaginal sonography in the diagnosis of adenomyosis: which findings are most accurate? Ultrasound Obstet Gynecol. 2007 Sep;30(3):341-5. doi: 10.1002/uog.3985. PMID 17659649
- [Background] Meredith SM, Sanchez-Ramos L, Kaunitz AM. Diagnostic accuracy of transvaginal sonography for the diagnosis of adenomyosis: systematic review and metaanalysis. Am J Obstet Gynecol. 2009 Jul;201(1):107.e1-6. doi: 10.1016/j.ajog.2009.03.021. Epub 2009 Apr 26. PMID 19398089
- [Background] Gordts S, Brosens JJ, Fusi L, Benagiano G, Brosens I. Uterine adenomyosis: a need for uniform terminology and consensus classification. Reprod Biomed Online. 2008 Aug;17(2):244-8. doi: 10.1016/s1472-6483(10)60201-5. PMID 18681999